CLINICAL TRIAL: NCT05175079
Title: A Randomised Controlled Trial On Effect Of Acupressure On Nausea And Vomiting In Women With Hyperemesis Gravidarum
Brief Title: Acupressure in Hyperemesis Gravidarum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FF-2017-195
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Hyperemesis Gravidarum
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accupressure group (Experimental): acupressure band apply to P6 (nei guan) point which located three fingers below the skin wrinkles of the anterior wrist.
  Acupressure band wear 3 times daily before breakfast, lunch and dinner for at least 10 minutes
  Interventions: Device: Acupressure band
- Control group (Placebo Comparator)
  Interventions: Other: Standard treatment hospital protocol

INTERVENTIONS:
Device: Acupressure band — acupressure band apply to P6 (nei guan) point which located three fingers below the skin wrinkles of the anterior wrist.
  Acupressure band wear 3 times daily before breakfast, lunch and dinner for at least 10 minutes
  Arms: Accupressure group
Other: Standard treatment hospital protocol — Intravenous metaclopromide 10mg PRN Intravenous fluids as per protocol
  Arms: Control group

SUMMARY:
To examine the degree of nausea, vomiting between the acupressure and control group in women with hyperemesis gravidarum

DETAILED DESCRIPTION:
A prospective RCT conducted at Department of Obst and Gynae, UKMMC. All pregnant women with a normal intrauterine pregnancy of ≤ 16 week gestation with hyperemesis gravidarum will be assessed by the medical officer/ specialist/ consultant in charge. Explanation regarding the research study will be given for patients who fulfill the inclusion and exclusion criteria. Patients who have understood the research study and consented will be recruited as subjects for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of vomiting before 16 weeks
2. Vomiting at least 2 times per day
3. Ketonuria on admission
4. Mid stream urine specimen that did not indicate infection

Exclusion Criteria:

1. Non viable pregnancy
2. Molar pregnancy
3. Overt clinical features of thyrotoxicosis
4. Known case of medical illness that associated with nausea and vomiting
5. Patient refusal or patients who are not able to give consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 90 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Degree of nausea and vomiting | day 1 to day 3
  measure the effect of acupressure using modified Pregnancy Unique Quantification of Emesis and Nausea (PUQE)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
No data are available for sharing

REFERENCES:
- [Derived] Mohd Nafiah NA, Chieng WK, Zainuddin AA, Chew KT, Kalok A, Abu MA, Ng BK, Mohamed Ismail NA, Nur Azurah AG. Effect of Acupressure at P6 on Nausea and Vomiting in Women with Hyperemesis Gravidarum: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Sep 1;19(17):10886. doi: 10.3390/ijerph191710886. PMID 36078602